CLINICAL TRIAL: NCT00423956
Title: Repair of Orthodontically-induced Tooth Root Resorption by Ultrasound in Human Subjects
Brief Title: Repair of Orthodontically-induced Tooth Root Resorption by Ultrasound
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Tarek El-Bialy, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6203
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Root Resorption
Keywords: Teeth root resorption, ultrasound, therapy
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sham Comparator (Sham Comparator): One side is experimental and the opposite side is Sham control.
  Interventions: Procedure: Repairing Induced tooth root resorption by ultrasound

INTERVENTIONS:
Procedure: Repairing Induced tooth root resorption by ultrasound — Repairing Induced tooth root resorption by ultrasound

SUMMARY:
Tooth-root resorption, also known as shortening or erosion,(TRR) is one of the adverse outcomes of dental trauma, orthodontic tooth movement and dental replantation/transplantation. Orthodontically induced inflammatory root resorption (OIIRR) is somewhat different from other types of TRR. The treatment protocol of teeth diagnosed with severe OIIRR or other forms of TRR always involves root canal treatment or extraction of these teeth in severe cases and prosthetic replacement. Sometimes teeth with minor TRR may stay for an extended period of time with compromised bite functions. Although several trials have been proposed to minimize or prevent TRR or OIIRR, none is capable of being used in clinical situation to treat TRR or OIIRR in humans except for Low Intensity Pulsed Ultrasound (LIPUS). However, research examining the use of LIPUS to treat OIIRR has been limited to simple orthodontic tooth tipping. In reality, tooth movement is a combination of different types of tooth movements, namely tipping, bodily, rotational, torque, intrusion and extrusion tooth movements. However, the literature have pointed out that torque tooth movement, especially when the root apices are torques against cortical plates of bone produces the most dramatic type of tooth root resorption with poor prognosis. Our long-term goal is to develop a standard protocol for treating severe tooth root resorption with poor prognosis in humans, regardless of origin. Our preliminary data demonstrates that LIPUS can produce healing of OIIRR in humans after simple tipping movement, this was confirmed by an in-vitro study on isolated cementoblasts. The objective of the present proposal is to evaluate the effect of different treatment protocols of LIPUS on the healing process of orthodontically induced tooth-root resorption due to torque (Complex)type of tooth movement in humans.

The study Hypotheses are (I) LIPUS treatment for 20 minutes per day for 4 weeks will be effective in repairing OIIRR due to torque tooth movement.

(II) The stimulatory effect of LIPUS to repair OIIRR due to torque tooth movement than LIPUS treatment is dose and time dependent.

DETAILED DESCRIPTION:
For each patient, specially designed springs will be used to achieve standard torque orthodontic tooth movement of the first premolars to induce OIIRR. The first molars will be stabilized, using a special appliance to help movement of the premolars. This type of appliance design has been used for many years in similar clinical trials by many researchers and has received wide acceptability without reported problems to the teeth during the experimental period. Ultrasound will be applied for twenty minutes per day, starting the day the springs are activated, for four weeks, using an ultrasound device (Exogen Inc., West Caldwell, NJ, USA). Only the first premolar will be receiving ultrasound. The patients will be instructed on how to have the ultrasound transducer. The non LIPUS treated premolars will be receiving sham transducers. A visual analogue scale will be provided to the patients to record any pain or discomfort that the patient might experience during or after application of ultrasound. It is expected that there will be no evidence of any deleterious effect on the intervening soft tissue as we did not informed with any discomfort experienced by the patients in our preliminary study. After four or eight weeks of LIPUS treatment, the springs will be removed, and the first premolars will be extracted, using a non-traumatic technique. The extracted teeth will be fixed, and studied by μ-CT then they will be processed to be analyzed histomorphometrically

ELIGIBILITY:
Inclusion Criteria:

* All the root apices of the experimental premolars should be completed.
* All experimental premolars should be sound and have no history of trauma/caries or root canal therapy.

Exclusion Criteria:

* Patients with incomplete experimental premolars' apices.
* 2- Any patient with experimental premolars that have a history of trauma/caries or root canal therapy.

Ages: 12 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of LIPUS on OITRR | Four weeks
Teeth Root length | four weeks
Root resorption lacunae number and volume | Four weeks

SECONDARY OUTCOMES:
Study the effect of LIPUS on alveolar bone remodeling | Four weeks
Rate of tooth movement | Rate of tooth movement at the time of extraction
  Teeth position before and after treatment will be measured to evaluate the possible effect of ultrasound on tooth movement.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tarek H El-Bialy, PhD, Study Chair — University of Alberta, Edmonton, AB, Canada
Locations (1):
- University of Alberta, Graduate Orthodontic program, Edmonton, Alberta, Canada